CLINICAL TRIAL: NCT01021072
Title: A Phase 1 Study of MABp1 in Patients With Advanced Cancers
Brief Title: A First in Man Study of MABp1 in Patients With Advanced Cancers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009-PT004
Record Dates: First submitted 2009-11-16; First posted 2009-11-26 (Estimated); Last update posted 2021-02-16 (Actual); Status verified 2021-02

CONDITIONS: Advanced Cancers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MTD (Experimental): The study will utilize a standard 3+3 design for dose escalation. Once the maximum tolerated dose has been reached, an expansion cohort, as well as tumor specific expansion cohorts will be explored.
  Interventions: Drug: MABp1

INTERVENTIONS:
Drug: MABp1 — 0.25 mg/kg,0.75 mg/kg,1.25 mg/kg, 3.75 mg/kg IV (in the vein) on day 1 of each 21 day cycle until progression or unacceptable toxicity develops.

SUMMARY:
The purpose of this study is to block interleukin-1 alpha activity with a True Human monoclonal antibody, thus interrupting the inflammatory response that supports tumor growth/metastasis and which drives the cachexic process.

An adaptive design will be employed which will allow for the exploration of different dosing regimens, as well as tumor types that show preliminary evidence of efficacy.

ELIGIBILITY:
Inclusion Criteria:

* pathologically confirmed advanced malignancy that is metastatic or unresectable and which is refractory to standard therapy or for which thee is no standard therapy that provides benefits for >/= 3 months
* measurable or non-measurable disease at baseline
* at least 4 weeks since the last dose of chemotherapy, radiation therapy, immunotherapy, or surgery; at least 6 weeks for therapy which is known to have delayed toxicity; at least 4 weeks since treatment with biologic/targeted therapies; at least 2 weeks since last hormonal therapy
* will not be treated with any other chemotherapy, immunotherapy, radiotherapy or investigational drug while enrolled on this protocol
* age >/= 18 year, male or female
* Eastern Cooperative Oncology Group performance status 0,1,or 2
* Serum potassium and magnesium levels within institutional normal limits. Total serum calcium or ionized calcium level must be greater than or equal to the low limit of normal.
* Adequate renal function, defined by serum creating </= 1.5 x ULN
* Adequate hepatic function
* Adequate bone marrow function WOCBP, a negative serum pregnancy test result at screening.
* WOCBP or men whose sexual partners are WOCBP who are willing to use an acceptable method of contraception for at least 1 month prior to study entry, for the duration of the study, and for at least 3 months after the last dose of study medication
* Signed and dated IRB approved ICF before any protocol specific screening procedures are performed

Exclusion Criteria:

* serious uncontrolled medical disorder or active infection which would impair the patient to receive protocol therapy.
* Uncontrolled or significant cardiovascular diseae
* dementia or altered mental status that would prohibit the understanding or rendering of informed consent
* not recovered from the adverse effects of prior therapy at the time of enrollment </= grade 1
* symptomatic brain metastases which are either untreated or uncontrolled by surgery and or radiotherapy
* received extensive prior radiation therapy to the bone marrow
* immunocompromised, including subjects know to be infected with HIV
* history of hypersensitivity to compounds of similar chemical or biologic composition to the antibody women how are pregnant or breastfeeding
* WOCBP or men whose sexual partners are WOCBP who are unwilling or unable to use an acceptable method of contraception for at least 1 month prior to study entry, for the duration of the study, and for at least 3 months after the last dose of study medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2010-03-31 (Actual); Primary Completion 2012-10-31 (Actual); Study Completion 2013-08-31 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose | one year

SECONDARY OUTCOMES:
Tumor response | one year
Cachexia Response | 8 weeks
  Change in LBT as measured by DEXA

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - M.D. Anderson Cancer Institute, Houston, Texas
  - MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Derived] Hong DS, Hui D, Bruera E, Janku F, Naing A, Falchook GS, Piha-Paul S, Wheler JJ, Fu S, Tsimberidou AM, Stecher M, Mohanty P, Simard J, Kurzrock R. MABp1, a first-in-class true human antibody targeting interleukin-1alpha in refractory cancers: an open-label, phase 1 dose-escalation and expansion study. Lancet Oncol. 2014 May;15(6):656-66. doi: 10.1016/S1470-2045(14)70155-X. Epub 2014 Apr 17. PMID 24746841